CLINICAL TRIAL: NCT07251153
Title: A Phase 1, Two Parts, Open-label, Pharmacokinetic Comparison of Vonafexor Acid and Its Lysine Salt (EYP651) in Healthy Volunteers and Evaluation of Potential Drug-Drug Interactions
Brief Title: Pharmacokinetic Comparison of Vonafexor Acid and Its Lysine Salt and Evaluation of Potential Drug-Drug Interactions
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Enyo Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EYP001-110; 2025-522915-40-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-14; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Healthy Adult Male and Female Volunteers
Keywords: Drug-Drug Interactions; Pharmacokinetic; Pharmacodynamic
MeSH Terms: interventions — Cytochrome P-450 CYP3A Inhibitors; Cytochrome P-450 CYP2C8

STUDY DESIGN:
Intervention Model Description: Crossover study model for the part A of the study. Parallel study model for the part B of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Vonafexor low dose (Experimental): Vonafexor low dose 1 tablet per day
  Interventions: Drug: EYP651/Vonafexor low dose
- Vonafexor high dose (Experimental): Vonafexor high dose 1 tablet per day
  Interventions: Drug: EYP651/Vonafexor high dose
- EYP651 low dose (Experimental): EYP651 low dose 1 tablet per day
  Interventions: Drug: EYP651/Vonafexor low dose
- EYP651 high dose (Experimental): Vonafexor high dose 1 tablet per day
  Interventions: Drug: EYP651/Vonafexor high dose; Drug: EYP651/CYP3A4 inhibitor; Drug: EYP651/Transporter substrate; Drug: EYP651/CYP2C8 and CYP2C9 substrate
- CYP3A4 inhibitor (Active Comparator): Oral daily administration
  Interventions: Drug: EYP651/CYP3A4 inhibitor
- Transporter substrate (Active Comparator): Oral daily administration
  Interventions: Drug: EYP651/Transporter substrate
- CYP2C8 and CYP2C9 substrate (Active Comparator): Oral daily administration
  Interventions: Drug: EYP651/CYP2C8 and CYP2C9 substrate

INTERVENTIONS:
Drug: EYP651/Vonafexor low dose — Repeated daily dosing with EYP651 or Vonafexor Acid for 5 days, cross-over at low dose according to period 1
  Arms: EYP651 low dose; Vonafexor low dose
Drug: EYP651/Vonafexor high dose — Repeated daily dosing with EYP651 or Vonafexor Acid for 5 days, cross-over at high dose according to period 1
  Arms: EYP651 high dose; Vonafexor high dose
Drug: EYP651/CYP3A4 inhibitor — Repeated daily dosing with EYP651 alone in period 1, and combined administration repeated daily dosing of EYP651 with index drug 1 (CYP3A4 inhibitor) in period 3. Parallel group 1
  Arms: CYP3A4 inhibitor; EYP651 high dose
Drug: EYP651/Transporter substrate — Repeated daily dosing with EYP651 alone in period 1, and combined administration repeated daily dosing of EYP651 with index drug 2 (Transporter substrate) in period 3. Parallel group 2
  Arms: EYP651 high dose; Transporter substrate
Drug: EYP651/CYP2C8 and CYP2C9 substrate — Repeated daily dosing with EYP651 alone in period 1, Repeated daily dosing with the index drug 3 alone in period 2 and combined administration repeated daily dosing of EYP651 with index drug 3 (CYP2C8 and CYP2C9 substrate) in period 3. Parallel group 3
  Arms: CYP2C8 and CYP2C9 substrate; EYP651 high dose

SUMMARY:
The purpose of this study is to define and compare the pharmacokinetic (PK) and pharmacodynamic (PD) profile of EYP651 at two dose levels and compare it with Vonafexor Acid PK and PD profile, the Part A.

In addition, Part B of the trial will assess the Drug-Drug Interactions (DDI) potential with the high dose of EYP651.

DETAILED DESCRIPTION:
The two parts are open-label and randomized, with a 2 periods, cross-over design for part A and a 3-period-parallel-arm design for Part B.

Expected duration for part A is approximately 8 weeks and Part B is approximately 12 weeks for each participating subject.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subject, aged 18-65 years inclusive.
* Females of childbearing potential: commitment to use a highly effective method of birth control which result in a low failure rate.

Females of non-childbearing potential: either at least 3 months surgically sterilized or at least 1-year postmenopausal confirmed by the follicle stimulating hormone (FSH) level.

Males: commitment to use an adequate contraceptive method consistently and correctly.

* Negative pregnancy test for childbearing potential women or FSH ≥ 40 IU/mL for postmenopausal women.
* Non-smoker subject or smoker of maximum 5 cigarettes a day and able to stop during the study.
* Body Mass Index (BMI) between 18 and 30 kg/m2 inclusive.
* Considered as healthy after a comprehensive clinical assessment (detailed medical history and complete physical examination).
* Normal Blood Pressure and Heart Rate.
* Normal ECG recording on a 12-lead ECG.
* Laboratory parameters within the normal range of the laboratory (hematology, hemostasis, blood chemistry tests, urinalysis).
* Normal dietary habits.
* Signing a written informed consent prior to selection.
* Covered by Health Insurance System and / or in compliance with the recommendations of National Law in force relating to biomedical research.

Exclusion Criteria:

* Any relevant history or presence of cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic, haematological, neurologic, psychiatric, systemic or infectious disease.
* Frequent headaches and / or migraine, recurrent nausea and / or vomiting.
* Symptomatic hypotension whatever the decrease of blood pressure or asymptomatic postural hypotension.
* Blood donation in the 2 months before administration.
* General anaesthesia in the 3 months before administration.
* Presence or history of drug allergic condition and/or hypersensitivity.
* Inability to abstain from intense muscular effort.
* Any drug intake (except paracetamol and contraceptives) during the month prior to the first administration.
* History or presence of drug or alcohol abuse (alcohol consumption > 40 grams / day).
* Excessive consumption of beverages with xanthine bases (> 4 cups or glasses / day).
* Positive Hepatitis B surface antigen or anti Hepatitis C Virus antibody, or positive results for Human Immunodeficiency Virus 1 or 2 tests.
* Positive results for drugs of abuse tests.
* No possibility of contact subject in case of emergency.
* Subject who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development.
* Exclusion period of a previous study.
* Administrative or legal supervision.
* Subject who would receive more than 6'000 euros as indemnities for his participation in biomedical research within the 12 last months, including the indemnities for the present study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2025-12-18 (Estimated); Study Completion 2026-10-28 (Estimated)

PRIMARY OUTCOMES:
Part A: Pharmacokinetic Area Under the Curve (AUC) | 1 day
  Compare the single dose PK AUC of EYP651 and Vonafexor
Part A: Pharmacokinetic Maximum Plasma Concentration (Cmax) | 1 day
  Compare the single dose PK Cmax of EYP651 and Vonafexor
Part A: Pharmacokinetic AUC | 5 days
  Compare the multiple dose PK AUC of EYP651 and Vonafexor
Part A: Pharmacokinetic Cmax | 5 days
  Compare the multiple dose PK Cmax of EYP651 and Vonafexor
Part B: CYP3A4 inhibition change in AUC | 5 days
  To assess the effect of strong CYP3A4 inhibition on the pharmacokinetic AUC of EYP651 using Index drug 1, to evaluate EYP651 as an object of CYP3A4 inhibition
Part B: CYP3A4 inhibition change in Cmax | 5 days
  To assess the effect of strong CYP3A4 inhibition on the pharmacokinetic Cmax of EYP651 using Index drug 1, to evaluate EYP651 as an object of CYP3A4 inhibition
Part B: Transporter sensitive substrate change in AUC | 5 days
  To characterize the effect of EYP651 on the pharmacokinetic AUC of transporter sensitive substrate (Index drug 2) with EYP651 as the precipitant
Part B: Transporter sensitive substrate change in Cmax | 5 days
  To characterize the effect of EYP651 on the pharmacokinetic Cmax of transporter sensitive substrate (Index drug 2) with EYP651 as the precipitant
Part B: CYP2C8/CYP2C9 sensitive substrate change in AUC | 5 days
  To characterize the effect of EYP651 on the pharmacokinetic AUC of CYP2C8/CYP2C9 sensitive substrate (Index drug 3) with EYP651 as the precipitant
Part B: CYP2C8/CYP2C9 sensitive substrate change in Cmax | 5 days
  To characterize the effect of EYP651 on the pharmacokinetic Cmax of CYP2C8/CYP2C9 sensitive substrate (Index drug 3) with EYP651 as the precipitant

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofins Optimed, Gières, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline published results might be shared upon request with researchers who provide a methodologically sound proposal and to achieve objectives as set in the approved proposal.
Time Frame: PD will be shared deidentified and from 3 months and ending 5 years following article publication.